CLINICAL TRIAL: NCT06735508
Title: An Exploratory Study of the Personalized MRNA Neoantigen Vaccine in Combination with Adebrelimab As Adjuvant Treatment for Patients with Resected Non-small Cell Lung Cancer
Brief Title: MRNA Neoantigen Vaccine in Non-Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: Shanghai Regenelead Therapies Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NSCLC-IIT-RGL
Record Dates: First submitted 2024-11-28; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-11

CONDITIONS: NSCLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm A (Experimental): Safe run-in phase and Dose Expansion phase
  Interventions: Drug: mRNA Neoantigen Vaccine; Drug: Adebrelimab

INTERVENTIONS:
Drug: mRNA Neoantigen Vaccine — mRNA Neoantigen Vaccine
Drug: Adebrelimab — Adebrelimab is a programmed death-ligand 1 antibody.

SUMMARY:
Brief Summary: This study is an open, prospective, exploratory clinical trial designed to evaluate the safety,ability, immunogenicity, and preliminary efficacy of a personalized neoantigen mRNA vaccine in combination with adebelimab as adjuvant treatment for patients with non-small cell lung cancer (NSCLC).

The primary objectives of this study are to answer the following key questions:

1. The incidence of dose-limiting toxicities (DLTs) during the designated observation period.
2. The incidence and severity of adverse events (AEs) and serious adverse events (SAEs).
3. The determination of the maximum tolerated dose (MTD) or maximum administered dose (MAD).

ELIGIBILITY:
Inclusion Criteria:

* Surgically resected and histologically or cytologically confirmed NSCLC according to the United States Joint Committee on Cancer (AJCC) eighth edition guidelines
* Qualify and sufficient tumor samples for genetic testing and neoantigen analysis
* There are no EGFR and ALK gene alteration
* Eastern Cooperative Oncology Group (ECOG) score of United States: 0 or 1 point
* Estimated survival ≥ 6 months
* Qualify and sufficient blood samples for immunogenicity and biomarkers before and after treatment, of which the blood samples for genetic testing during the screening period must be free of blood transfusions, blood products and other hematopoietic stimulating factors within 7 days before collection
* Postoperative complications have recovered, or complications are lower than Clavien-Dindo complication grade 3
* There was no evidence of disease in clinical examination, chest and abdomen contrast-enhanced CT and baseline radiological evaluation of head MRI within 14 days before the first dose
* Female subjects of childbearing potential must have a serum pregnancy test within 7 days prior to the first dose with a negative result; and must be non-lactating
* Female subjects of childbearing potential and male subjects whose partners are women of childbearing potential must agree to comply with contraceptive requirements from the time of signing the informed consent form until 90 days after the end of the last treatment (see "Contraceptive methods" in Annex V for details)

Exclusion Criteria:

* Histologically or cytologically diagnosed small cell lung cancer (SCLC), or mixed tumors with small cell components, or neuroendocrine tumors or sarcomatoid carcinomas with large cell components
* Any person who is not suitable for immunotherapy as assessed by the investigator
* Presence of autoimmune diseases, except for hypothyroidism due to autoimmune thyroiditis that only requires hormone replacement therapy
* Evidence of active tuberculosis infection within 1 year prior to initiation of study treatment, regardless of treatment
* Subjects with a known history of interstitial pneumonia or a high suspicion of interstitial pneumonia, or evidence of active interstitial pneumonia on chest CT during the pre-screening period; Known history of idiopathic pulmonary fibrosis, history of organizing pneumonia (such as bronchiolitis obliterans or cryptogenic organizing pneumonia); and subjects who may interfere with the detection or management of suspected drug-related pulmonary toxicity
* Severe infection (such as intravenous infusion of antibiotics, antifungal or antiviral drugs required according to clinical diagnosis and treatment standards) within 28 days before starting study treatment, or active infection that has received therapeutic intravenous or oral antibiotics within 14 days before starting study treatment
* Known allergy to the study drug or any of its excipients, or history of severe allergic reactions to other vaccines
* Subject has a history of other malignancies within the past 5 years or at the same time, excluding cured carcinoma in situ of the cervix, basal cell carcinoma of the skin or squamous cell carcinoma of the skin, localized prostate cancer after radical resection, ductal carcinoma in situ after radical resection (hormonal therapy for non-metastatic prostate cancer or breast cancer is allowed), and papillary thyroid carcinoma
* Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation
* Patients with congenital or acquired immunodeficiency, such as cellular immunodeficiency (e.g., DiGeorge syndrome, T-negative severe combined immunodeficiency [SSCID]) or combined T-cell and B-cell immunodeficiency (e.g., T- and B-negative combined immunodeficiency, Wiskott-Aldrich syndrome, ataxia telangiectasia, common variable immunodeficiency); or human immunodeficiency virus (HIV) infection
* Active hepatitis B (defined as a positive active hepatitis B virus surface antigen [HBsAg] test result during the screening period with detection of HBV DNA ≥500IU/mL or above the upper limit of normal for the study center), or hepatitis C (defined as a positive hepatitis C antibody [HCV-Ab] test result and HCV-RNA positive during the screening period)
* Has poorly controlled or severe cardiovascular disease, such as severe/unstable angina, symptomatic congestive heart failure (NYHA Class III. or IV.), myocardial infarction within 6 months prior to initiation of study treatment, or unstable angina pectoris within 1 month prior to initiation of study treatment, or presence of cardiac arrhythmias requiring treatment or intervention, or poorly controlled hypertension (systolic blood pressure ≥ 150mmHg, diastolic blood pressure ≥90mmHg) after adequate treatment
* In the opinion of the investigator, the subject has a history of other serious systemic diseases, or other reasons are not suitable for participating in this clinical study (such as any other disease that may affect the subject's compliance with the study treatment, interfere with the interpretation of the study results, or expose the subject to safety risks, or the tumor tissue sequencing data analysis results show that there are not enough neoantigens available for vaccine preparation, or the vaccine preparation fails); Other circumstances judged by the investigator that may affect the conduct of clinical research and the judgment of research results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
safety and tolerability | From the start of study treatments until 30 days after last dose of study treatments.
  Percentage of subjects who meet the criteria of DLT in DLT observation period
MTD or MAD | From the start of study treatments until the end of the safety run-in phase, about 4 months.
  Determine the maximum tolerated dose (MTD) or maximum administered dose (MAD) and recommended expansion dose (RDE) of mRNA Neoantigen in combination with adebelimab in the adjuvant treatment of resectable NSCLC after surgery

SECONDARY OUTCOMES:
immunogenicity | From the sugery til the end of study treatment，about 18 months.
  Change in immunogenicity compared to baseline, rate of the immune response
Preliminary efficacy | 3years
  DFS rate and OS rate at 18 months/24 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No